CLINICAL TRIAL: NCT00658398
Title: Effect of an Interactive Computer Program to Prevent Alcohol Misuse. A Multicentre Randomized Controlled Trial. The BREVALCO Study.
Brief Title: The BREVALCO Study, Effect of an Interactive Computer Program to Prevent Alcohol Misuse
Acronym: BREVALCO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P060252
Record Dates: First submitted 2008-04-09; First posted 2008-04-15 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2013-08

CONDITIONS: AOD Misuse
Keywords: Alcohol; dependency
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICP to prevent alcohol misuse. (Experimental): Interactive Computer Program (ICP) to prevent alcohol misuse.
  Interventions: Behavioral: Interactive Computer Program to prevent alcohol misuse.
- ICP to enhance balanced diet (Sham Comparator): 2. Interactive Computer Program to enhance balanced diet (sham intervention)
  Interventions: Behavioral: Interactive Computer Program to prevent alcohol misuse.

INTERVENTIONS:
Behavioral: Interactive Computer Program to prevent alcohol misuse. — Interactive Computer Program with questionnaires, video and informations

SUMMARY:
The purpose of this study is to evaluate the effect of a brief computer program to prevent alcohol misuse for patients consulting in an emergency department and screened for alcohol misuse.

DETAILED DESCRIPTION:
Purpose: to evaluate the effect of a brief computer program to prevent alcohol misuse for patients consulting in an emergency department and screened for alcohol misuse.

Design: A randomized controlled trial with patients blinded of study hypotheses. Randomization will be stratified on centers and the sex

Interventions:

Patients randomized in the experimental group will participate in an interactive computer program with video, questionnaires and information related to alcohol misuse. They will also be contacted by phone at 1 month and 3 months to reinforce the effect of the intervention.

Patients randomized in the control group will participate in an interactive computer program with questionnaires and information related to healthy diet. They will also be contacted by phone at 1 month and 3 months to reinforce the effect of the intervention.

Participants: all patients consulting in an emergency department will be screened regarding their alcohol consumption and misuse. All patients screened as having alcohol misuse will be invited to participate in the trial.

Outcomes: the main outcome is the declared alcohol consumption at 12 months. Patients will be evaluated by phone at 3, 6 and 12 months by an independent outcome assessor.

Analyses: An intention to treat analyses will be performed Number of patients: 600 patients will be included Number of centers:3 centres (university hospital) will participate

ELIGIBILITY:
Inclusion Criteria:

* age >=18
* patients consulting in an emergency department
* screened for alcohol misuse or dependence (i.e. for women: AUDIT score>5 or consumption of more than 14 alcohol drinks per week For men: AUDIT score>8 or consumption of more than 7 alcohol drinks per week)
* informed and signed consent form
* clinical exam performed
* having social protection

Exclusion Criteria:

* vital risk
* patients having mental disorder,
* patient unable to answer the questions and to participate in the computer program because of their clinical condition
* patients no understanding French languages
* patient already being treated for alcohol disorder
* patients asking for a specific treatment for their alcohol disorder
* patients unable to answer to the follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2008-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The mean number of alcohol drinks by day in the previous week, at 12months. | 12 months

SECONDARY OUTCOMES:
the AUDIT score (0-40) at 12 months, | 12 months
the DSM-IV-TR criteria of alcohol abuse or dependence at 12 months | 12 months
the mean number of drunkenness or alcohol intoxications with behaviour problems per day in the previous week at 12 months, | 12 months
Three numerical scales of social satisfaction (0 to 10) based on health, family life or relationship, occupation or daily activity at 12 months, | 12 months
the percentage of consultations at an ED at 12 months, | 12 months
the percentage of consultations at hospital at 12 months, | 12 months
the rate of acceptance of a long-term follow-up | 12 months
the rate of suicide attempts. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michel LEJOYEUX, PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe hospitalier Bichat Claude Bernard, Paris, France